CLINICAL TRIAL: NCT04924309
Title: Stress in Couples Undergoing Assisted Reproduction Technology With Donor Insemination and Its Impact on Reproductive Outcomes
Brief Title: Stress in Couples Undergoing Assisted Reproduction Technology With Donor Sperm and Its Impact on Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20210328
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing assisted reproductive technology with donor sperm
  Interventions: Other: Exposure: donor sperm
- Patients undergoing assisted reproductive technology with husband's semen due to male factor

INTERVENTIONS:
Other: Exposure: donor sperm — One group use donor sperm through the process of assisted reproduction and the other uses husband's semen.
  Groups: Patients undergoing assisted reproductive technology with donor sperm

SUMMARY:
Donor sperm provides a viable option for patients with significant male factor infertility. However, since the source of sperm is not from the male partner, the psychological burden of these couples is more pronounced and complex than other patients.The purpose of this study is to investigate the stress faced by participants undergoing assisted reproduction with donor sperm and to further investigate its impact on pregnancy outcomes.

DETAILED DESCRIPTION:
The number of infertility patients has increased significantly in recent years, and infertility caused by the male partner accounts for about 30%-50% of infertility factors. Donor sperm provides a viable option for patients with significant male factor infertility. However, since the source of sperm is not from the male partner, the psychological burden of these couples is more pronounced and complex than other patients. Many factors such as social, marital, and family problems may contribute to their depressed emotional state. And the impact of these negative emotions on pregnancy outcomes cannot be ignored. In this study, investigators intend to investigate the stress faced by participants undergoing assisted reproduction with donor sperm to provide a reliable basis for future psychological interventions and health education for this group of patients and improve the quality of life of infertility patients.

ELIGIBILITY:
Inclusion Criteria:

* Female partners' >18< 40 years
* Male partners' >18< 40 years
* Patients undergoing assisted reproductive technology with donor sperm or husband's semen due to male factor

Exclusion Criteria:

* Female partners with polycystic ovary
* Female partners with insufficiency or premature ovarian failure
* Female partners with endometriosis
* Female partners with abnormal profile of thyroid hormones
* Chromosomal abnormalities of either spouse
* Mental disorder of either spouse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing assisted reproductive technology with donor sperm or husband's semen due to male factor
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 8 months
  Implantation rate is defined as number of sacs per embryo transferred.
clinical pregnancy rate | 8 months
  presence of at least one gestational sac on ultrasound of 6 weeks

SECONDARY OUTCOMES:
fertilization rate | 8 months
  No. of fertilized oocyte divided by No. of inseminated cumulus-oocyte complexes (COCs)
cleavage rate | 8 months
  No. of cleaved embryo divided by No. of fertilized oocyte
Total gonadotropin use | 8 months
  Total gonadotropin use of each participant
Ovarian hyperstimulation syndrome (OHSS) rates | 8 months
  OHSS rates in both study groups
Number of oocytes retrieved | 8 months
Metaphase II (MII) oocytes | 8 months
  the number of mature oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Zhu, Study Chair — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China